CLINICAL TRIAL: NCT02968407
Title: Peer- and Self-rating of Open Surgery Skills Using Objective Structured Assessment of Technical Skills
Brief Title: Peer- and Self-rating of Open Surgery Skills
Acronym: self-rate
Status: Completed | Type: Observational
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Diana Haunstrup Bregner Overgaard, Research Scholar, Copenhagen Academy for Medical Education and Simulation
Other Study IDs: H-16031885
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Peer- and self-rating — Participants will be given a print and a e-mail of the modified OSATS global rating scale and will be introduced to how the rating scale is used to rate technical performance. The participant will receive a USB stick each allowing the participant to see a video of his/her own performance and two videos from previous post-test performances from participants enrolled in the course. One video is a video of a participant who performed poorly,the other is from a participant who performed well. The participants will be asked to watch and rate the videos of their peers' performance first and afterwards watch and rate the participants own video performance. The investigators choose to let the participants rate their peers' performances before their own, so the participants will have the best opportunities to self-rate. Participants will be asked to email the results of their ratings to the principal investigator within 3 days. And expert in surgery will also rate the videos using OSATS.

SUMMARY:
The study group want to investigate whether doctors, who are in the beginning of their training to become surgeons, can rate themself and their peers using Objective Structured Assessment of Technical Skills. Participants have participated in a 6 weeks course in basic open surgical skills. At the end of the course the participants will be examined at at videotaped test. The participants will be asked to rate their own video and two videos of other trainees' performances. Ratings will be compared to expert ratings.

DETAILED DESCRIPTION:
The study is a prospective, descriptive study investigating whether doctors are able to rate their own and their peers' performance in a basic open surgery skill course. At the end of the course in basic open surgery, participants will be examined at the post-test as described in the protocol "The effect of group dynamics in surgical skill training". After the participants complete the post-test, participants will be asked to participate in this additional study. The participants will receive no instructions on this additional study, before they complete the study "The effect of group dynamics in surgical skill training".

ELIGIBILITY:
Inclusion Criteria:

* Participants are medical doctors and medical students who completed the study "The effect of group dynamics in surgical skill training" as part of the control group.
* The participants must be willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Participants who do not finish the basic open surgery course
* Medical doctors and medical students enrolled in the study "The effect of group dynamics in surgical skill training" that are randomized to dyad training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Setting The participants will follow the basic open surgery skill course as described in the protocol "The effect of group dynamics in surgical skill training".
  Participants Participants are medical doctors and medical students who completed the study "The effect of group dynamics in surgical skill training" as part of the control group.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Differences between the participants' rating score of his/her own performance and the experts' rating score of the participants' performance | six months
  To investigate whether medical doctors are able to rate their own performance in a basic open surgery skill course using a modified OSATS rating scale

SECONDARY OUTCOMES:
Differences between the participants' rating score of his/her peers performances and experts' rating score of the peers' performances | six months
  To investigate whether medical doctors are able to rate their peers' performance in a basic open surgery skill course using a modified OSATS rating scale
Differences in the correlation of self-rating score and expert rating score between participants who are rated in the upper quartile by experts compared to participants who are rated in the lower quartile by experts | Six months
  To investigate the correlation between level of competency and the ability to self-rate in a basic open surgery skill course using a modified OSATS rating scale
Differences in the correlation of participants' rating scores and experts' rating scores between participants first and second rating of their peers performance. | six months
  To investigate whether there is progression in the participants ability to rate their peers performances using OSATS

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the data within the study group
Supporting Information: Study Protocol
Time Frame: Expected to be published during 2018